CLINICAL TRIAL: NCT07001215
Title: Effect of CPAP Versus APAP in Patients With Obesity Undergoing Bariatric Surgery Protocol
Acronym: ObesAOS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Ramon y Cajal (Other)
Collaborators: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Principal Investigator, Laura Pozuelo Sánchez, University Diploma in Nursing from UAM and Bachelor's Degree in Psychology from UNED. Biomedical researcher at IRYCIS., Hospital Universitario Ramon y Cajal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 111/25
Record Dates: First submitted 2025-05-22; First posted 2025-06-03 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-05

CONDITIONS: Sleep Apnea, Obstructive; Bariatric Surgery; Obesity; Treatment Adherence and Compliance; Continuous Positive Airway Pressure (CPAP)
Keywords: Obstructive Sleep Apnea (OSA); Continuous Positive Airway Pressure (CPAP); Automatic Positive Airway Pressure (APAP); Bariatric Surgery; Obesity
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity; Treatment Adherence and Compliance | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: Single-center, randomized, parallel-group, open-label, controlled clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- APAP Group (Experimental): APAP Group: They will receive treatment with AutoCPAP. The device automatically adjusts the air pressure according to the patient's needs, and usage data and respiratory events will be manually collected at each visit.
  Interventions: Device: In the intervention group, patients will be treated with auto-adjusting APAP, providing variable pressures throughout the sleep hours.
- CPAP group (Active Comparator): CPAP Group: They will receive treatment with conventional CPAP. The device will provide a fixed and constant air pressure, and follow-up will be conducted through in-person visits and titration with APAP after adherence to verify the optimal pressure. The initial CPAP pressure will be individually calculated using Hoffstein's formula based on parameters such as body mass index (BMI), neck circumference, and apnea-hypopnea index (AHI).
  Interventions: Device: CPAP

INTERVENTIONS:
Device: In the intervention group, patients will be treated with auto-adjusting APAP, providing variable pressures throughout the sleep hours. — AutoCPAP will be prescribed to patients undergoing bariatric surgery.
  Other Names: APAP; Automatic Positive Airway Pressure
  Arms: APAP Group
Device: CPAP — In the control group, patients will be treated with CPAP.
  Other Names: Continuous Positive Airway Pressure
  Arms: CPAP group

SUMMARY:
Introduction Obstructive sleep apnea (OSA) is a common disorder in obese patients, especially those undergoing bariatric surgery. OSA is characterized by upper airway obstruction during sleep, leading to intermittent hypoxia and sleep fragmentation. Obesity and OSA are closely related conditions that can exacerbate each other. Positive airway pressure therapy is essential for managing OSA, but adherence to therapy can be challenging, particularly in patients who experience rapid physiological changes after bariatric surgery.

Objective This study aims to determine whether automatic positive airway pressure therapy (APAP) improves nightly usage hours compared to continuous positive airway pressure therapy (CPAP) in obese patients undergoing bariatric surgery. Secondary objectives include evaluating the percentage of nights with therapy use over 4 hours, reduction of the residual apnea-hypopnea index (AHI), changes in daytime sleepiness, pressure requirements, side effects, sleep-related quality of life, reduction in in-person visits, and optimization of healthcare resources.

Methodology A randomized, parallel-group, open-label, controlled clinical trial will be conducted. Adult patients eligible for bariatric surgery with a diagnosis of moderate to severe OSA (AHI > 15) requiring positive pressure therapy will be included. Participants will be randomized to receive either APAP or CPAP. Follow-up will be conducted over 12 months after surgery, with assessments at 3, 6, and 12 months. Data will be collected on treatment adherence, residual AHI, OSA symptoms, daytime sleepiness, quality of life, and treatment costs.

APAP therapy is expected to improve nightly usage hours compared to CPAP. It is also expected that APAP will show better adaptation to changing pressure needs after bariatric surgery. Data will be analyzed to evaluate the effectiveness and cost-efficiency of both therapies.

This study will provide evidence on the efficacy of APAP compared to CPAP in obese patients undergoing bariatric surgery. The results will help optimize the treatment of OSA in this population and improve patients' quality of life. Additionally, the study is expected to contribute to the optimization of healthcare resources by reducing in-person visits and repeated sleep studies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 to 80 years who meet the criteria for bariatric surgery and are on the surgical waiting list after approval by the bariatric surgery committee (BMI ≥35, or BMI ≥30 with comorbidities).
* Diagnosis of moderate or severe sleep apnea, defined by an Apnea-Hypopnea Index (AHI) >15, requiring treatment according to protocol ("Patients with an AHI of 15 or higher will be treated with CPAP if they have hypertension, excessive daytime sleepiness, or sleep-related symptoms not explained by other causes" [17]).
* Patients must be able to read and understand the informed consent and provide signed consent.

Exclusion Criteria:

* Patients with central sleep apnea or periodic breathing
* Patients with any active neoplasm
* Patients with severe uncontrolled psychiatric disorders, alcoholism, or active drug addiction
* Patients with unacceptable surgical/anesthetic risk
* Patients who have undergone previous surgery for OSA or who have been treated with positive airway pressure and did not tolerate it

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-09-15 (Estimated); Study Completion 2028-09-15 (Estimated)

PRIMARY OUTCOMES:
APAP vs. CPAP: Impact on Nightly Usage in Obese Patients Undergoing Bariatric Surgery | Obese patients undergoing bariatric surgery will be evaluated during the 3 months prior to surgery and at 3, 6, and 12 months postoperatively in patients with OSA undergoing bariatric surgery.
  To determine whether APAP therapy increases nightly usage hours compared to CPAP therapy in obese patients undergoing bariatric surgery. Unit of Measure: Average hours of PAP use per night (measured via device data).

SECONDARY OUTCOMES:
Therapy Adherence Over Time | 3 months before bariatric surgery and at 3, 6, and 12 months postoperatively.
  To measure and compare the percentage of nights with therapy usage exceeding 4 hours in both groups (APAP and fixed CPAP). Unit of Measure: Percentage of nights with ≥4 hours of PAP use.
Reduction in Residual AHI | 3 months before bariatric surgery and at 3, 6, and 12 months postoperatively.
  To evaluate the reduction in the residual Apnea-Hypopnea Index (AHI) in both groups. Unit of Measure: Residual AHI (events per hour).
Daytime Sleepiness | 3, 6, and 12 months postoperatively
  To assess changes in daytime sleepiness using validated scales (e.g., Epworth Sleepiness Scale) in both groups. Unit of Measure: Total ESS score (range: 0-24; higher scores indicate greater sleepiness).
Pressure Requirement Trends | (3 months pre-surgery and 3, 6, and 12 months postoperatively).
  To evaluate and compare changes in positive airway pressure (PAP) requirements, measured in cm H₂O, in patients treated with APAP or CPAP over time.
  Unit of Measure: Pressure level (cm H₂O).
Pressure Adaptability of APAP | 3, 6, and 12 months postoperatively
  To assess the adaptability of APAP therapy to varying pressure requirements over time, compared to fixed-pressure CPAP, in patients with OSA following bariatric surgery.
  Unit of Measure: Variability in delivered pressure (cm H₂O).
Side Effects Monitoring | (3 months pre-surgery and 3, 6, and 12 months postoperatively).
  To measure and compare the presence of side effects (e.g., nasal dryness, skin irritation) in both groups. Unit of Measure: Incidence of reported side effects (percentage of patients affected).
Sleep Quality (assessed using the Pittsburgh Sleep Quality Index) | (3 months pre-surgery and 3, 6, and 12 months postoperatively).
  To assess sleep quality using the validated Pittsburgh Sleep Quality Index (PSQI) questionnaire.in both groups. Unit of Measure: Total PSQI score (range: 0-21; higher scores indicate poorer sleep quality).
General Quality of Life (assessed using the EuroQol-5D) | 3 months pre-surgery and 3, 6, and 12 months postoperatively.
  To assess general quality of life using the validated EuroQol-5D (EQ-5D) questionnaire. Unit of Measure: EQ-5D Utility Index and Visual Analogue Scale (VAS) score 0-100.
Reduction in Outpatient Visits | (3 months pre-surgery and 3, 6, and 12 months postoperatively).
  To analyze the potential reduction in outpatient clinic visits in the APAP group compared to the CPAP group. Unit of Measure: Number of outpatient visits per patient.
Healthcare Resource Optimization | (3 months pre-surgery and 3, 6, and 12 months postoperatively).
  To evaluate the reduction in repeated sleep studies as an indicator of healthcare resource optimization in patients treated with APAP compared to CPAP.
  Unit of Measure: Number of repeated sleep studies per patient.
STOP-BANG Questionnaire Accuracy | (3 months pre-surgery and 3, 6, and 12 months postoperatively).
  To assess the sensitivity and specificity of the STOP-BANG questionnaire for detecting OSA in bariatric patients, and to determine whether a new cutoff point is needed to optimize its performance in this population. Unit of Measure: STOP-BANG total score (range 0 to 8); sensitivity and specificity percentages for different cutoff points.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Pozuelo-Sánchez, Nurse, Principal Investigator — Iricys
Locations (1):
- Hospital Universitario Ramón y Cajal,, Madrid, Spain, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kermelly SB, Lajoie AC, Boucher ME, Series F. Impact of continuous positive airway pressure mode on adherence to treatment in obstructive sleep apnea patients awaiting bariatric surgery. J Sleep Res. 2021 Oct;30(5):e13288. doi: 10.1111/jsr.13288. Epub 2021 Feb 6. PMID 33547713
- [Background] Katasani T, Holt G, Al-Khyatt W, Idris I. Peri- and Postoperative Outcomes for Obstructive Sleep Apnoea Patients after Bariatric Surgery-a Systematic Review and Meta-analysis. Obes Surg. 2023 Jul;33(7):2016-2024. doi: 10.1007/s11695-023-06557-8. Epub 2023 May 4. PMID 37140722
- [Background] Collen J, Lettieri CJ, Eliasson A. Postoperative CPAP use impacts long-term weight loss following bariatric surgery. J Clin Sleep Med. 2015 Mar 15;11(3):213-7. doi: 10.5664/jcsm.4528. PMID 25515283
- [Background] de Raaff CAL, de Vries N, van Wagensveld BA. Obstructive sleep apnea and bariatric surgical guidelines: summary and update. Curr Opin Anaesthesiol. 2018 Feb;31(1):104-109. doi: 10.1097/ACO.0000000000000542. PMID 29176373
- [Background] Joosten SA, Hamilton GS, Naughton MT. Impact of Weight Loss Management in OSA. Chest. 2017 Jul;152(1):194-203. doi: 10.1016/j.chest.2017.01.027. Epub 2017 Feb 6. PMID 28185772
- [Background] Kapur VK, Auckley DH, Chowdhuri S, Kuhlmann DC, Mehra R, Ramar K, Harrod CG. Clinical Practice Guideline for Diagnostic Testing for Adult Obstructive Sleep Apnea: An American Academy of Sleep Medicine Clinical Practice Guideline. J Clin Sleep Med. 2017 Mar 15;13(3):479-504. doi: 10.5664/jcsm.6506. PMID 28162150
- [Background] Xu YX, Wang SS, Wan YH, Su PY, Tao FB, Sun Y. Association of sleep fragmentation with general and abdominal obesity: a population-based longitudinal study. Int J Obes (Lond). 2024 Sep;48(9):1258-1265. doi: 10.1038/s41366-024-01547-x. Epub 2024 May 28. PMID 38806646
- [Background] Mediano O, Gonzalez Mangado N, Montserrat JM, Alonso-Alvarez ML, Almendros I, Alonso-Fernandez A, Barbe F, Borsini E, Caballero-Eraso C, Cano-Pumarega I, de Carlos Villafranca F, Carmona-Bernal C, Carrillo Alduenda JL, Chiner E, Cordero Guevara JA, de Manuel L, Duran-Cantolla J, Farre R, Franceschini C, Gaig C, Garcia Ramos P, Garcia-Rio F, Garmendia O, Gomez Garcia T, Gonzalez Pondal S, Hoyo Rodrigo MB, Lecube A, Madrid JA, Maniegas Lozano L, Martinez Carrasco JL, Masa JF, Masdeu Margalef MJ, Mayos Perez M, Mirabet Lis E, Monasterio C, Navarro Soriano N, Olea de la Fuente E, Plaza G, Puertas Cuesta FJ, Rabec C, Resano P, Rigau D, Roncero A, Ruiz C, Salord N, Saltijeral A, Sampol Rubio G, Sanchez Quiroga MA, Sans Capdevila O, Teixeira C, Tinahones Madueno F, Maria Togeiro S, Troncoso Acevedo MF, Vargas Ramirez LK, Winck J, Zabala Urionaguena N, Egea C; el Spanish Sleep Network. International Consensus Document on Obstructive Sleep Apnea. Arch Bronconeumol. 2022 Jan;58(1):52-68. doi: 10.1016/j.arbres.2021.03.017. Epub 2021 Mar 24. English, Spanish. PMID 33875282
- [Background] Young T, Palta M, Dempsey J, Skatrud J, Weber S, Badr S. The occurrence of sleep-disordered breathing among middle-aged adults. N Engl J Med. 1993 Apr 29;328(17):1230-5. doi: 10.1056/NEJM199304293281704. PMID 8464434